CLINICAL TRIAL: NCT03803761
Title: A Phase 2 Study of Copanlisib (BAY 80-6946) in Combination With Fulvestrant in Patients With Metastatic Breast Cancer Progressing After Aromatase Inhibitor Plus CDK 4/6 Inhibitor
Brief Title: A Study of a New Drug Combination, Copanlisib and Fulvestrant, in Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00048; NCI-2019-00048 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI10195; 10195 (Other: Duke University - Duke Cancer Institute LAO); 10195 (Other: CTEP); UM1CA186704 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-01-15 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Malignant Neoplasm in the Brain; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — copanlisib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (copanlisib, fulvestrant) (Experimental): Patients receive copanlisib IV over 1 hour on days 1, 8, and 15 and fulvestrant IM over 1-2 minutes on days 1 and 15 of cycle 1 and on day 1 beginning cycle 2. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Copanlisib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Copanlisib — Given IV
  Other Names: BAY 80-6946; PI3K Inhibitor BAY 80-6946
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238

SUMMARY:
This phase I/II trial studies the side effects and how well copanlisib works when given together with fulvestrant in treating patients with estrogen receptor positive (ER+) and human epidermal growth factor receptor 2 negative (HER2-) breast cancer that has spread to other places in the body (advanced) and progressing after prior treatment. HER2 and ER are two types of proteins called receptors that can affect the growth of breast cancer cells. Additionally, investigators hope to learn from this study if tumor genetic information is important for predicting whether this type of breast cancer will respond to fulvestrant and copanlisib. Copanlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Hormone therapy using fulvestrant may fight breast cancer by blocking the use of estrogen by the tumor cells. Giving copanlisib and fulvestrant may work better in treating patients with ER+ and HER2- breast cancer compared to fulvestrant alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish safety of the combination of copanlisib and fulvestrant (FC). II. Evaluate the response rate (RR) of the combination of copanlisib and fulvestrant in patients with estrogen-receptor positive (ER+)/human epidermal growth factor receptor 2 (HER2) negative metastatic breast cancer that has previously progressed on aromatase inhibitor (AI)/cyclin dependent kinase (CDK) 4/6 inhibitor therapy.

SECONDARY OBJECTIVES:

I. Estimate progression-free survival (PFS) in patients treated with copanlisib and fulvestrant stratifying by actionable PIK3CA mutation, actionable PIK3CA or PTEN mutation, or wild type PIK3CA and PTEN.

II. Estimate the RR in subjects with PTEN loss by immunohistochemistry (IHC) analysis performed retrospectively.

III. Evaluate toxicity in patients treated with FC in Phase II.

EXPLORATORY OBJECTIVES:

I. Evaluate copanlisib pharmacokinetics (PK) when given in combination with fulvestrant.

II. Explore association between intrinsic subtype and response to FC therapy. III. Assess baseline levels and treatment-induced proteomic changes and correlate with response to FC.

IV. Evaluate circulating tumor deoxyribonucleic acid (DNA) (ctDNA) mutations at baseline and over time for response predictors at baseline, clonal evolution associated with treatment, and resistance mechanisms at disease progression.

V. Evaluate PFS in patients with baseline ctDNA PIK3CA actionable mutations versus (vs.) those with wild type PK3CA.

VI. To evaluate genomic and gene expression changes in tumor cells and in associated tumor microenvironment before and after administration of copanlisib in combination with fulvestrant and at the time of progression.

VII. Evaluate circulating markers of metabolism before and after PI3K inhibitor therapy which may predict treatment response and resistance mechanisms.

OUTLINE:

Patients receive copanlisib intravenously (IV) over 1 hour on days 1, 8, and 15 and fulvestrant intramuscularly (IM) over 1-2 minutes on days 1 and 15 of cycle 1 and on day 1 beginning cycle 2. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with estrogen receptor positive (ER+), human epidermal growth factor receptor 2 (HER2) negative metastatic breast cancer (MBC) who have progressed on combination therapy with an aromatase inhibitor and cyclin-dependent kinase 4/6 (CDK 4/6) inhibitor

  * Note: Postmenopausal females are considered of childbearing potential unless they are surgically or permanently sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. Documentation of postmenopausal status must be provided
* Measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST1.1)
* Patients must have had tumor sequencing for evaluation of actionable PIK3CA or PTEN mutations performed in a Clinical Laboratory Improvement Act (CLIA) certified, College of American Pathologist (CAP) tested and bioinformatics-validated testing lab PRIOR to enrollment in this current protocol. If available patient tumor sequencing status must be provided to University of North Carolina (UNC) principal investigator (PI) at consent, and prior to any additional screening procedures. The testing may have been done at any time prior to enrollment. For patients who have not yet had tumor genomic assessment, after consultation with the PI, tumor specimens will be sent to the UNC Hospitals Clinical Molecular Genetics Laboratory for assessment of the Solid Tumor Mutation Panel. In this case, results of genetic testing by the UNC lab must be available prior to the first on study disease assessment (i.e., prior to day 1 of cycle 4). In this case, the study will cover the cost of the Solid Tumor Panel
* Female subjects who are not of childbearing potential

  * Note: Because no dosing or adverse event data are currently available on the use of copanlisib in combination with fulvestrant in patients <18 years of age, and only postmenopausal women with ER+/HER2 negative MBC are eligible or appropriate for treatment with fulvestrant, children and pregnant or pre-menopausal women are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* No prior treatment history with fulvestrant or a PI3K inhibitor
* Subject has not received more than 2 prior lines of chemotherapy in the metastatic setting
* Subject must have washout period from prior systemic anti-cancer therapy of at least 21 days (or 5 half-lives of the systemic anti-cancer therapy, whichever is shorter) before the start of study treatment
* Subject must have washout period from prior radiation therapy of at least 2 weeks before the start of study treatment
* Subjects with a history of brain metastases are allowed if they are not on steroid therapy and there is no evidence of intracranial disease progression symptomatically or by imaging within 28 days prior to study registration
* Hemoglobin >= 9.0 g/dL (collected no more than 7 days before starting treatment)
* Leukocytes >= 3,000/mcL (collected no more than 7 days before starting treatment)
* Absolute neutrophil count >= 1,500/mcL (collected no more than 7 days before starting treatment)
* Platelets >= 100,000/mcL (collected no more than 7 days before starting treatment)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (collected no more than 7 days before starting treatment) (< 3 x ULN for patients with Gilbert syndrome, patients with cholestasis due to compressive adenopathies of the hepatic hilum or documented liver involvement)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN) OR =< 5 x institutional ULN if liver metastases present (collected no more than 7 days before starting treatment)
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2 (collected no more than 7 days before starting treatment)
* Fasting blood glucose < 120 mg/dL (collected no more than 7 days before starting treatment)
* Lipase =< 1.5 x ULN (collected no more than 7 days before starting treatment)
* International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x ULN (collected no more than 7 days before starting treatment)
* Left ventricular ejection fraction (LVEF) >= 50%
* Subject must agree to provide archival tumor material for research and/or agree to undergo a tumor biopsy for research if the tumor is accessible for biopsy prior to study treatment
* Ability to understand and the willingness to comply with study procedures and to sign a written informed consent document
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial

Exclusion Criteria:

* Previous assignment to treatment during this study. Patients permanently withdrawn from study participation will not be allowed to re-enter the study
* Concomitant participation in another clinical study with investigational medicinal product
* Subjects who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Immunosuppressive therapy is not allowed while on study
* Subjects who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to copanlisib, fulvestrant, or PI3K inhibitors
* Subjects with moderate or severe hepatic impairment (ie, Child-Pugh B or C)
* Copanlisib is primarily metabolized by CYP3A4. Therefore, the concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and strong inducers of CYP3A4 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) are not permitted from 14 days prior to enrollment until the end of the study. Other medications that are prohibited while on copanlisib treatment:

  * Herbal medications/preparations (except for vitamins)
  * Anti-arrhythmic therapy other than beta blockers or digoxin
* Systemic corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not permitted while on study. Previous corticosteroid therapy must be stopped or reduced to the allowed dose at least 7 days prior to the computed tomography (CT)/magnetic resonance imaging (MRI) screening; if a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose before the screening; patients may be using topical or inhaled corticosteroids; short-term (up to 7 days) systemic corticosteroids above 15 mg prednisolone or equivalent will be allowed for the management of acute conditions (e.g., treatment non-infectious pneumonitis); the use of corticosteroids as antiemetics prior to copanlisib administration will not be allowed
* Uncontrolled intercurrent illness, including but not limited to, psychiatric illness/social situations that would limit compliance with study requirements
* Major surgical procedure or significant traumatic injury (as judged by the investigator) within 28 days prior to start of treatment, or not recovered from major side effects, or open biopsy within 7 days before start of study treatment
* Patients with non-healing wound, ulcer, or bone fracture not due to breast cancer
* Patients with active, clinically serious infections > grade 2 (Common Terminology Criteria for Adverse Events [CTCAE] version [v]5.0)
* Patients with glycosylated hemoglobin (HbA1c) > 8.5% at screening
* Proteinuria of >= CTCAE grade 3 as assessed by a 24 hour (h) protein quantification or estimated by urine protein: creatinine ratio > 3.5 on a random urine sample
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication
* Congestive heart failure > New York Heart Association (NYHA) class 2

  * Note: Class III NYHA Heart failure classification: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain
  * Note: Class IV NYHA Heart failure classification: Patients with cardiac disease resulting in the inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.

Other cardiovascular-related abnormalities or therapy that prohibit study participation are:

* Myocardial infarction less than 6 months before start of study medications
* Unstable angina (angina symptoms at rest), new onset angina (begun within the last 3 months)
* Uncontrolled arterial hypertension despite optimal medical management
* Anti-arrhythmic therapy (exceptions: beta blockers or digoxin are permitted)

  * Pregnant or lactating (Pregnant women or women who are breastfeeding are excluded from this study because copanlisib is a PI3K inhibitor agent with the potential for teratogenic or abortifacient effects; there is no safety data in pregnancy; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with copanlisib, breastfeeding should be discontinued if the mother is treated with copanlisib and/or fulvestrant; fulvestrant may also cause fetal harm and based on animal studies, may impair fertility in females of reproductive potential)
  * Hepatitis B virus (HBV) or hepatitis C virus (HCV). All patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus lab panel; patients positive for hepatitis B virus surface antigen (HBsAg) and/or hepatitis B virus core antibody (HBcAb) will be eligible if they are negative for deoxyribonucleic acid (DNA), these patients should receive prophylactic antiviral therapy; patients positive for anti-HCV antibody will be eligible if they are negative for HCV ribonucleic acid (RNA)
  * Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral agents that are strong CYP3A4 inhibitors or inducers and who are unwilling or unable to change to antiretroviral therapies without such interactions are ineligible because of the potential for pharmacokinetic interactions with copanlisib
  * Subjects with seizure disorder requiring medication
  * Subjects with evidence or history of bleeding diathesis; any hemorrhage or bleeding event >= CTCAE grade 3 within 4 weeks prior to the start of study medication
  * Blood or platelet transfusion less than 7 days before start of study treatment or myeloid growth factors within 14 days prior to treatment
  * History of concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
  * History of, or current autoimmune disease
  * Concurrent diagnosis of pheochromocytoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-13 (Estimated); Primary Completion 2022-02-19 (Estimated); Study Completion 2022-02-19 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 30 days post treatment
  Toxicities will be tabulated based on type and grade.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From start of treatment to time of progression or death, assessed up to 30 days post treatment
  PFS will be estimated using the Kaplan Meier method, with median and 95% confidence interval (CI) reported.
Response rate | Up to 30 days post treatment
  Response rate will be reported for subjects with PTEN loss by immunohistochemistry (IHC) analysis performed retrospectively. This will be done across cohorts.
Incidence of adverse events | Up to 30 days post treatment
  Toxicities will be tabulated based on type and grade. Any toxicity seen in more than 10% of patients will be reported, and all grade 3-4 toxicities will be reported.

OTHER OUTCOMES:
Pharmacokinetics (PK) and pharmacodynamic data (RPPA) | Up to 30 days post treatment
  Descriptive statistics will be provided.
Biomarkers analysis | Up to 30 days post treatment
  Prognostic effect of biomarker for PFS will be examined by the Kaplan Meier (KM) method or/and Cox proportional hazard model and for objective response rate (ORR) using logistic regression model. Predictive effect of biomarker will be explored by examining the interaction effect of biomarker and arm in Cox or logistic regression model. For markers measured along multiple time points, generalized linear mixed effects model will be used to model longitudinal trajectories along time with the inference focus on the arm factor, without and with adjustment for other covariates. Two sample t-test or Wilcoxon rank sum test will be applied to compare time-matched biomarkers between the two arms or two patient subsets. Paired sample t-test or Wilcoxon signed rank test will be applied to compare subject-specific biomarkers between two time points. Multiple comparisons will be adjusted to control false discovery rate. Proposed subset analyses will be applicable to biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Dees, Principal Investigator — Duke University - Duke Cancer Institute LAO
Locations (7):
- United States (7):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - NYP/Weill Cornell Medical Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Texas Medical Branch, Galveston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm